CLINICAL TRIAL: NCT03286491
Title: Development of Clinical Decision Support System to Define 30 Day Adverse Clinical Events (Non Fatal Myocardial Infarction, Cardiac Related Death or Coronary Intervention) for Patients Presenting to Emergency Department With Acute Coronary Syndrome
Brief Title: Clinical Decision Support System to Define 30 Day Adverse Clinical Events for Emergency Department Acute Coronary Syndromes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turkish Ministry of Health Izmir Teaching Hospital (Other Government)
Responsible Party: Principal Investigator, Serhat Akay, M.D., Turkish Ministry of Health Izmir Teaching Hospital
Other Study IDs: TurkishMOHITH
Record Dates: First submitted 2017-09-15; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Acute Coronary Syndrome; Clinical Decision Support System
Keywords: acute coronary syndrome, risk classification, 30 day adverse event, clinical decision support system
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients presenting with acute coronary syndrome: Patients presenting to emergency department with acute coronary syndrome
  Interventions: Diagnostic Test: Further cardiac imaging

INTERVENTIONS:
Diagnostic Test: Further cardiac imaging — Study patients will be reviewed whether they will have coronary interventions in 30 days

SUMMARY:
Acute coronary syndromes are among main complains for patients presenting to emergency department. Risk classification systems are used to classify patients to appropriate risks and help physicians manage diagnosis strategies and treatments. Purpose of this study is to develop a clinical decision support system for patients presenting to emergency department with the help of statistical machine learning.

DETAILED DESCRIPTION:
Acute coronary syndromes are among main complains for patients presenting to emergency department and create a burden to emergency departments and hospitals. Risk classification systems were developed and used to classify patients to appropriate risk groups. According to risk classification, different diagnosis and treatment modalities can be used and help physicians manage diagnosis strategies and treatments. Purpose of this study is to develop a clinical decision support system for patients presenting to emergency department with the help of statistical machine learning.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to emergency department with acute chest pain consistent with acute coronary syndrome

Exclusion Criteria:

* Patients with less than 18 years old
* Patients presenting with ST-segment elevation myocardial infarction
* Patients presenting with other causes of acute chest pain (pneumothorax, pulmonary -embolism, aortic dissection
* Decline to participate in study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting to emergency deparmtent with acute chest pain consistent with acute coronary syndrome will be included for analysis.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-08-12 (Actual); Primary Completion 2017-12-12 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
Non fatal myocardial infarction, cardiac related death or coronary intervention in 30 days | 30 days
  Patients will be screened for 30 days for Non fatal myocardial infarction, cardiac related death or coronary intervention (coronary angiogram, coronary artery bypass surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No